CLINICAL TRIAL: NCT06986044
Title: EVALUATION OF SALIVA AND SERUM HEME OXYGENASE, ARYLESTERASE AND NUCLEAR FACTOR ERYTHROID 2-RELATED FACTOR 2 LEVELS IN PATIENTS WITH STAGE III PERIODONTITIS
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Zeynep Hazan YILDIZ, Doctor, Saglik Bilimleri Universitesi
Other Study IDs: GülhaneDiş
Record Dates: First submitted 2025-04-22; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Health; Periodontitis Stage III
Keywords: total antioxidan status; total oxidan status; oxidative stress index; arylesterase; heme oxygenase; nuclear factor erythroid 2 related factor 2; saliva; serum; stage III periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- stage III grade B periodontitis: Pocket deep ≤ 6 mm, clinical attachment loss ≥ 5 mm, tooth loss related to periodontitis ≤ 4, radiographic bone loss/age between 0.25-1 and periodontal tissue destruction compatible with biofilm accumulation.
  Interventions: Diagnostic Test: Serum Total Oxidant Status; Diagnostic Test: Salivary Total Oxidant Status; Diagnostic Test: Serum Total Antioxidant Status; Diagnostic Test: Salivary Total Antioxidant Status; Diagnostic Test: Serum Oxidative Stress Index; Diagnostic Test: Salivary Oxidative Stress Index; Diagnostic Test: Serum Arylesterase; Diagnostic Test: Salivary Arylesterase; Diagnostic Test: Serum Heme Oxygenase; Diagnostic Test: Salivary Heme Oxygenase; Diagnostic Test: Serum Nuclear Factor Erythroid 2 Related Factor 2; Diagnostic Test: Salivary Nuclear Factor Erythroid 2 Related Factor 2; Diagnostic Test: Gingival Index; Diagnostic Test: Plaque Index; Diagnostic Test: Bleeding on Probing Index; Diagnostic Test: Clinical Attachment Loss; Diagnostic Test: Pocket Deep
- periodontally health: Pocket deep ≤ 3 mm, bleeding on probing index ≤ %10 and gingival index ≤ 1
  Interventions: Diagnostic Test: Serum Total Oxidant Status; Diagnostic Test: Salivary Total Oxidant Status; Diagnostic Test: Serum Total Antioxidant Status; Diagnostic Test: Salivary Total Antioxidant Status; Diagnostic Test: Serum Oxidative Stress Index; Diagnostic Test: Salivary Oxidative Stress Index; Diagnostic Test: Serum Arylesterase; Diagnostic Test: Salivary Arylesterase; Diagnostic Test: Serum Heme Oxygenase; Diagnostic Test: Salivary Heme Oxygenase; Diagnostic Test: Serum Nuclear Factor Erythroid 2 Related Factor 2; Diagnostic Test: Salivary Nuclear Factor Erythroid 2 Related Factor 2; Diagnostic Test: Gingival Index; Diagnostic Test: Plaque Index; Diagnostic Test: Bleeding on Probing Index; Diagnostic Test: Clinical Attachment Loss; Diagnostic Test: Pocket Deep

INTERVENTIONS:
Diagnostic Test: Serum Total Oxidant Status — Serum total oxidant status
Diagnostic Test: Salivary Total Oxidant Status — Salivary Total Oxidant Status
Diagnostic Test: Serum Total Antioxidant Status — Serum Total Antioxidant Status
Diagnostic Test: Salivary Total Antioxidant Status — Salivary Total Antioxidant Status
Diagnostic Test: Serum Oxidative Stress Index — Serum Oxidative Stress Index
Diagnostic Test: Salivary Oxidative Stress Index — Salivary Oxidative Stress Index
Diagnostic Test: Serum Arylesterase — Serum Arylesterase
Diagnostic Test: Salivary Arylesterase — Salivary Arylesterase
Diagnostic Test: Serum Heme Oxygenase — Serum Heme Oxygenase
Diagnostic Test: Salivary Heme Oxygenase — Salivary Heme Oxygenase
Diagnostic Test: Serum Nuclear Factor Erythroid 2 Related Factor 2 — Serum Nuclear Factor Erythroid 2 Related Factor 2
Diagnostic Test: Salivary Nuclear Factor Erythroid 2 Related Factor 2 — Salivary Nuclear Factor Erythroid 2 Related Factor 2
Diagnostic Test: Gingival Index — Gingival Index
Diagnostic Test: Plaque Index — Plaque Index
Diagnostic Test: Bleeding on Probing Index — Bleeding on Probing Index
Diagnostic Test: Clinical Attachment Loss — Clinical Attachment Loss
Diagnostic Test: Pocket Deep — Pocket Deep

SUMMARY:
Periodontal disease is a chronic and progressive inflammatory disease in which the hard and soft tissues that support the teeth are damaged. It is caused by the interaction between harmful bacteria and the body's immune responses, and most periodontal tissues are damaged by the body's abnormal response to these microorganisms and their products. When bacteria enter the body, immune cells (neutrophils) produce reactive oxygen species (ROS) in a process called the "respiratory burst". These ROS damage cells, causing tissue destruction through a variety of mechanisms, including DNA damage, fat oxidation and protein damage. Studies have shown that neutrophils from individuals with periodontal disease produce more ROS than neutrophils from healthy individuals. High amounts of ROS lead to oxidative damage to gum tissue, periodontal ligament and alveolar bone. Oxidative stress occurs when antioxidants in the body are insufficient or when high levels of ROS are present. Therefore, disruption of the balance between oxidant and antioxidant activities is considered an important cause of oxidative damage in periodontal tissues. Parameters such as total antioxidant status (TAS), total oxidant status (TOS) and oxidative stress index (OSI) are used to determine oxidative stress.

Furthermore, some enzymes such as arylesterase (ARE), heme oxygenase (HO) and nuclear factor erythroid 2-related factor 2 (NRF-2) are involved in defense mechanisms against oxidative stress. Many recent studies have shown a strong association between oxidative stress and periodontal disease.

DETAILED DESCRIPTION:
This study was divided into 2 groups, 37 systemically and periodontally health individuals and 37 systemically healthy individuals with stage III grade B periodontitis were included. Clinical periodontal parameters plaque index (PI), gingival index (GI), probing pocket depth (SCD), bleeding on probing (BOP) and clinical attachment level (CAL) were recorded and saliva and serum samples were collected. ELISA method was used for analyses of TOS, TAS, OSI, ARE, HO-1, NRF-2 levels.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* between the ages of 18-65

Exclusion Criteria:

* Patients with systemic diseases and/or conditions that may affect periodontal tissues (cardiovascular diseases, immune system diseases, rheumatoid arthritis, diabetes mellitus, chemotherapy/radiotherapy).
* taking any medication that may have an effect on periodontal tissues,
* less than 20 natural teeth excluding third molars
* used antibiotics, anti-inflammatory or immunosuppressive drugs
* periodontal treatment in the last 6 months
* smokers
* pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: periodontally healthy 19 female and 18 male subjects with a mean age of 39.48 years.
  periodontitis state III individuals, 20 females and 17 males with a mean age of 39.05 years.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
serum and saliva TAS (mmol Trolox Eq/L) levels | 6 months
  TAS concentrations were evaluated utilizing an innovative automated colorimetric assay, originally developed by Erel. The outcomes were reported as millimoles of Trolox equivalent per liter (mmol Trolox Eq/L).
  Total antioxidant levels are significantly lower in periodontitis patients compared to healthy individuals, suggesting increased oxidative stress associated with periodontal inflammation.
serum and saliva TOS (µmol H₂O₂ Eq/L) levels | 6 months
  TOS concentrations were determined through a distinct automated colorimetric technique, also described by Erel. Results were expressed as micromoles of hydrogen peroxide equivalent per liter (µmol H₂O₂ Eq/L). Compared to healthy controls, periodontitis patients show higher total oxidant levels, which may contribute to tissue destruction and disease progression.
serum and saliva OSI levels | 6 months
  TAS values (initially in mmol Trolox Eq/L) were converted to µmol Trolox Eq/L. OSI was then computed using the following formula: OSI = [(TOS, µmol/L) / (TAS, µmol Trolox Eq/L)] × 100.
  The oxidative stress index is significantly higher in periodontitis patients compared to healthy individuals, reflecting an imbalance between oxidants and antioxidants.
serum and saliva ARE (U/L) levels | 6 months
  Arylesterase activity was assessed using commercially available assay kits (Rel Assay Diagnostics, Turkey). For the measurement of arylesterase activity, phenylacetate was used as the substrate. The enzymatic activity was calculated based on the molar extinction coefficient of the phenol formed (1,310 M-¹cm-¹). One unit of arylesterase activity was defined as the amount of enzyme required to hydrolyze 1 µmol of phenol per minute under the assay conditions and was also expressed as U/L. Arylesterase activity is significantly decreased in periodontitis patients compared to healthy controls, suggesting impaired antioxidant enzyme function.
serum and saliva NRF-2 (ng/ml) levels | 6 months
  The level of NRF-2 was quantified using an enzyme-linked immunosorbent assay (ELISA) kit (BT lab.). In this assay, wells were pre-coated with human NRF-2-specific antibodies. Samples containing NRF2 were added to the wells, allowing target binding. Subsequently, a biotin-conjugated anti-NRF-2 antibody was applied, followed by streptavidin-horseradish peroxidase (HRP) conjugate. After washing to remove unbound components, a substrate solution was added, producing a colorimetric reaction proportional to the amount of NRF-2 present. The reaction was terminated by adding an acidic stop solution, and absorbance was measured at 450 nm. It is suggested that the reduced expression of NRF-2 in periodontitis patients, relative to healthy controls, contributes to increased oxidative stress and tissue damage.
serum and saliva HO-1(ng/ml) levels | 6 months
  The concentration of HO-1 was measured using an ELISA kit (BT Lab.) Wells were pre-coated with human HO-1-specific antibodies. Following the addition of samples, human HO-1 proteins bound to the immobilized antibodies. A biotinylated anti-HO-1 antibody and subsequently streptavidin-HRP conjugate were introduced. After removal of unbound components via washing, a substrate solution was added to initiate color development, which was proportional to the HO-1 concentration. The reaction was stopped using an acidic solution, and absorbance was recorded at 450 nm. Compared to healthy subjects, HO-1 is considered to be less expressed in periodontitis patients, potentially compromising antioxidant and anti-inflammatory defenses

SECONDARY OUTCOMES:
Gingival Index (GI) | 6 months
  Gingival Index (GI) (Löe ve Silness) : The presence of gingival inflammation was determined on 4 surfaces of all teeth using the GI score defined by Löe and Silness. The periodontal probe was moved over the tooth and index values between 0-3 were determined for each tooth. Compared to healthy individuals, a high gingival index score is frequently observed in periodontitis patients, indicating greater gingival inflammation.
Plaque Index (PI) | 6 months
  The presence of plaque and the Silness and Löe plaque index (PI) were obtained from 4 surfaces of the teeth after drying the teeth and index values between 0-3 were given. Plaque accumulation, as reflected by higher plaque index scores, is more prominent in periodontitis patients than in healthy controls.
Bleeding on Probing Index (BoP) | 6 months
  Bleeding in probing was evaluated as (+) if there was bleeding in the relevant area within 30 seconds after applying pressure to the gingival sulcus with the periodontal probe in 4 regions of all teeth with the weight of the probe itself, and as (-) if there was no bleeding. Compared to healthy controls, periodontitis patients demonstrate a higher incidence of bleeding on probing, indicating active inflammation and compromised periodontal tissue integrity.
Clinical Attachment Loss (CAL) (millimeter) | 6 months
  The distance between the cementoenamel junction of the tooth and the base of the periodontal pocket is calibrated millimetrically, with the clinical attachment level on 6 surfaces of all teeth. using a Williams periodontal probe. Clinical attachment level is significantly increased in periodontitis patients compared to healthy individuals, indicating the extent of periodontal tissue destruction.
Pocket Depth (PD) (millimeter) | 6 months
  Probing pocket depth was performed on 6 surfaces of all teeth using a millimetrically calibrated Williams periodontal probe. The distance of the free gingival margin to the pocket bottom was measured in millimeters. The probe was held parallel to the long axis and the force applied to the probe was released when resistance was encountered during the measurement. Probing pocket depth is significantly greater in periodontitis patients compared to healthy individuals, reflecting deeper periodontal pockets due to tissue destruction.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi Gülhane Diş Hekimliği Fakültesi, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided